CLINICAL TRIAL: NCT05508256
Title: CAtheter-Based Ablation of Atrial Fibrillation Compared to Conventional Treatment in Patients With Heart Failure With Preserved Ejection Fraction
Acronym: CABA-HFPEF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Kompetenznetz Vorhofflimmern e.V. (AFNET) (Unknown); Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Abdul Parwani, Head of Electrophysiology, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABA-HFPEF-DZHK27
Record Dates: First submitted 2022-08-10; First posted 2022-08-19 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mildly Reduced Ejection Fraction
Keywords: atrial fibrillation; heart failure; catheter ablation; medial therapy
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure

STUDY DESIGN:
Intervention Model Description: The CABA-HFPEF is an investigator-initiated, prospective, parallel-group, randomized, open, blinded endpoint assessment, interventional multicenter strategy trial. CABA-HFPEF compares two treatment strategies that employ established therapies within their approved indications.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter Ablation (Active Comparator): Symptomatic HFmrEF or HFpEF patients with AF that meet I/E criteria will be randomized 1:1 to receive either CA or usual medical care without the aim of CA. Patients assigned to rhythm control group will be treated with catheter ablation as first line therapy to restore and maintain sinus rhythm, additionally to the therapeutic recommendations of the current ESC guidelines for the management of atrial fibrillation (AF) and the current ESC Heart Failure (HF) guidelines.
  Interventions: Device: CE-marked Catheter Ablation
- Usual Medical Care (No Intervention): Symptomatic HFmrEF or HFpEF patients with AF that meet I/E criteria will be randomized 1:1 to receive either CA or usual medical care without the aim of CA. Subjects randomized to usual care will be treated according to current ESC guidelines for the management of AF and current ESC HF guidelines. Usual care of AF in the context of CABA-HFPEF consists of an initial treatment limited to rate control in addition to adequate antithrombotic therapy, typically oral anticoagulation.

INTERVENTIONS:
Device: CE-marked Catheter Ablation — Once patients have been randomized to the catheter ablation (CA) group, the ablation procedure must be performed within 4 weeks. CA will initially aim at pulmonary vein isolation.
  Arms: Catheter Ablation

SUMMARY:
The objective of CABA-HFPEF is to test whether catheter ablation (CA) for atrial fibrillation (AF) can prevent adverse cardiovascular outcomes in patients with heart failure with preserved (HFpEF) or mildly reduced ejection fraction (HFmrEF).

DETAILED DESCRIPTION:
HFpEF accounts for approximately half of HF diagnoses and HFmrEF adds another 20%. HFpEF patients are predisposed to AF with a prevalence of AF up to 65%. Conversely, the presence of AF increases the likelihood of subsequent HFpEF by up to 4-fold across diverse populations. The vulnerable hemodynamic state in HFpEF patients due to LV diastolic dysfunction can be significantly affected by AF with loss of atrial contraction and reduction in cardiac output. Thus, presence of AF in HFpEF patients leads to a significant increase in hospitalization, mortality and stroke.

Restoring and maintaining sinus rhythm in patients with HFpEF and AF could reduce cardiovascular (CV) outcomes. Catheter ablation (CA), particularly when performed as initial rhythm control, results in less recurrences of AF than anti arrhythmic drug therapy. In patients with HF with reduced ejection fraction (HFrEF) and AF, CA showed a significant reduction in all-cause mortality and worsening HF admissions compared to medical therapy.

No randomized clinical trial has tested or is currently testing the effects of CA on CV outcomes in patients with HFmrEF or HFpEF and AF. To address this, CABA-HFPEF tests whether CA can improve CV outcomes compared to usual care in these patients. The results of CABA-HFPEF will critically extend the current evidence on ablation-based rhythm control to this large population in dire need for treatments that improve clinical outcomes.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Age ≥18 years
2. Signed written informed consent
3. Clinical evidence of symptomatic heart failure (NYHA Class II-III)
4. Paroxysmal or persistent atrial fibrillation (less than 24 months after first diagnosis, documented at least on one 12-lead ECG)
5. Left ventricular ejection fraction (LVEF) 40-49%

   OR

   LVEF ≥ 50% with at least one of the following HFpEF echocardiography findings (any local measurement made during the screening epoch):

   A. LA enlargement defined by at least 1 of the following: LA width (diameter) ≥3.8 cm or LA length ≥5.0 cm or LA area ≥20 cm2 or LA volume ≥55 ml or LA volume index ≥29 ml/m2

   B. Left ventricular hypertrophy (septal thickness or posterior wall thickness ≥1.1 cm or relative wall thickness >0.42)
6. Patients with at least 1 of the following:

A. HF hospitalization (defined as HF listed as the major reason for hospitalization) within 6 months prior to screening visit and NT-proBNP >200 pg/ml for patients in sinus rhythm (SR) or >600 pg/ml for patients in AF at the time of blood sampling

B. NT-proBNP >300 pg/ml for patients in SR or >900 pg/ml for patients in AF on screening ECG

EXCLUSION CRITERIA:

1. Patient is unable or unwilling to provide infomed consent
2. Patient is not suitable for rhythm control of AF
3. Previous left atrial CA or surgical therapy of AF
4. Acutely decompensated HF, NYHA IV (patients can be enrolled after stabilization)
5. Valvular heart disease needing interventional or surgical treatment within 3 months
6. Heart surgery planned within 3 months
7. Prior heart transplant or listed for heart transplant or cardiac assist device implantation
8. Untreated hypothyroidism or hyperthyroidism (after successful treatment of thyroid dysfunction, patients may be enrolled)
9. Patient has absolute contra-indication to oral anticoagulation
10. Any disease that limits life expectancy to less than 1 year
11. Active systemic infection (after successful treatment of infection, patients may be enrolled)
12. Women currently pregnant or breastfeeding or women of childbearing potential without highly effective contraception (PEARL-Index < 1%)
13. Patient is included in another clinical trial
14. Inability to comply with the study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1548 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is defined as a composite of cardiovascular death, stroke and total (first and recurrent) unplanned cardiovascular hospitalization for heart failure or acute coronary syndrome. | Estimated first patient in to last patient out 48 months.

SECONDARY OUTCOMES:
All-cause mortality | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Cardiovascular death | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Stroke | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Total (first and recurrent) unplanned cardiovascular hospitalization for heart failure or acute coronary syndrome | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Unplanned hospitalization for atrial arrhythmia | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Total (first and recurrent) planned and unplanned cardiovascular hospitalizations | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Nights spent in hospital | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Days alive and out of hospital | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Atrial fibrillation burden (percentage of AF at 12 months FU Holter ECG) | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Change in left ventricular ejection fraction at 12 months FU | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Change in NYHA class at 12 months FU | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Change in EHRA score at 12 months FU | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months
Change in quality of life at 12 months FU | The secondary endpoints will be documented for at least 12 months following randomization. Estimated first patient in to last patient out 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Parwani, Dr., Principal Investigator — Head of Electrophysiology; Charité University Medicine Berlin, CVK; Paulus Kirchhof, Prof. Dr., Study Chair — Director Department of Cardiology, Heart and Vascular Center University Hamburg Eppendorf; Stefan Kääb, Prof. Dr., Study Chair — Department of Cardiology, Ludwig-Maximilians-University Hospital Munich; Tim Friede, Prof. Dr., Study Chair — Departement of Medical Statistics, University Medical Center Göttingen; Roland Tilz, Prof. Dr., Study Chair — Head of Electrophysiology Department, University Hospital Lübeck; Burkert Pieske, Prof. Dr., Study Chair — Independent
Locations (1):
- Charité University Medicine Berlin, Campus Virchow Klinikum, Berlin, Germany